CLINICAL TRIAL: NCT00364936
Title: Proposal to Create a Flagship Neurology and Palliative Care Service for South London
Brief Title: Development and Evaluation of a New Palliative Care Service for People Severely Affected With Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Prof I Higginson - Prinical investigator responsible, King's College London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS Society 676/01
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: palliative care; hospice; end-of-life; symptom control; evaluation; effectiveness
MeSH Terms: conditions — Multiple Sclerosis; Death | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Palliative care service

SUMMARY:
The primary purpose of this study is to develop, implement and conduct a preliminary evaluation of a new service for people who are severely affected by multiple sclerosis. The investigators conducted open interviews with patients, families and staff, plus a literature review to model and pilot this new service. Then the investigators developed, tested and ran the service and will evaluate it using a randomised controlled trial, where people affected by MS are randomised to either receive the service immediately (fast track group) or after a three month wait (standard best practice). This methodology follows that of the Medical Research Council (MRC) framework for the development and evaluation of complex services and treatments. The investigators interview people and their carers in the fast track and standard practice groups, and followed them over time. This phase of trial enables us to calculate sample size and test proof of concept for a full randomised trial. However, our working hypothesis was that there would be no difference between those people who received the fast track service or the standard best practice in terms of symptom controlled, and carer needs.

DETAILED DESCRIPTION:
Palliative care has been proposed to help meet the needs of patients who suffer progressive non-cancer conditions but this has not been tested. Multiple sclerosis is a chronic disease affecting the central nervous system affecting over 2.5 million people worldwide, and is the commonest cause of neurological disability in adults under 60 years. It is associated with a wide spectrum of physical symptoms, including loss of function of legs, arms and in many instances bladder and bowel dysfunction, pain, spasms, swallowing and communication and cognitive difficulties, many of which are as severe as among patients with cancer. Therefore it seems appropriate to try to develop palliative care services for this group of patients.

Our design followed the MRC Framework for the Evaluation of Complex Interventions. The investigators modelled a new palliative care and neurology service for patients affected by Multiple Sclerosis (MS) by conducting qualitative interviews with patients, families and staff, plus a literature review to model and pilot the service. Then the investigators started to offer the service and designed a delayed intervention randomised controlled trial to test its effectiveness as part of phase II of the MRC framework. Inclusion criteria for the trial were patients identified by referring clinicians as having unresolved symptoms or psychological concerns. A disability of scoring greater than 8 on the Expanded Disability Scale was identified as a benchmark. Consenting patients newly referred to the new service were randomised to either receive the palliative care service immediately (fast-track) or after a 12-week wait (standard best practice). Face to face interviews were conducted at baseline (before intervention), and at 4-6, 10-12 (before intervention for the standard-practice group), 16-18 and 22-24 weeks with patients and their carers using standard questionnaires to assess symptoms, palliative care outcomes, function, service use and open comments. The investigators choice of outcomes was based on a systematic literature review of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* Living in South East London
* Having possible palliative care needs. Referrers were encouraged to identify people as severely affected with MS based on their clinical need, rather than relying on any standardised measures of disability. However, since a large Canadian population study identified that approximately 15% of people with MS have an Expanded Disability Scale Score of 8 or more (out of a possible 10)23, this was also suggested to referrers as a benchmark for disability that would prompt consideration of referral. Examples of palliative care needs were given as unresolved symptoms, psychosocial concerns, and end of life issues, progressive illness or complex needs.

Exclusion Criteria:

* patients deemed as having urgent needs (following independent review by a consultant in palliative medicine) because of rapid deterioration or severe symptoms - these were seen immediately by the service.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Palliative Care Outcome Scale - Symptoms | 12 weeks

SECONDARY OUTCOMES:
Self-reported quality of life | 12 weeks
Impact of MS | 12 weeks
Psychosocial palliative care outcomes | 12 weeks
use of health and social services | 12 weeks
Experience of hospital services | 12 weeks
Carer burden and satisfaction | 12 weeks
Costs (formal and informal) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Polly Edmonds, FRCP, Principal Investigator — King's College Hospital / King's College London; Irene J Higginson, BMBS FRCP FFPHM PhD, Study Chair — King's College London
Locations (1):
- King's College Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Gruenewald DA, Higginson IJ, Vivat B, Edmonds P, Burman RE. Quality of life measures for the palliative care of people severely affected by multiple sclerosis: a systematic review. Mult Scler. 2004 Dec;10(6):690-704. doi: 10.1191/1352458504ms1116rr. PMID 15584496
- [Background] Edmonds P, Vivat B, Burman R, Silber E, Higginson IJ. 'Fighting for everything': service experiences of people severely affected by multiple sclerosis. Mult Scler. 2007 Jun;13(5):660-7. doi: 10.1177/1352458506071789. Epub 2007 Feb 9. PMID 17548447
- [Background] Edmonds P, Vivat B, Burman R, Silber E, Higginson IJ. Loss and change: experiences of people severely affected by multiple sclerosis. Palliat Med. 2007 Mar;21(2):101-7. doi: 10.1177/0269216307076333. PMID 17344258
- [Background] Higginson IJ, Vivat B, Silber E, Saleem T, Burman R, Hart S, Edmonds P. Study protocol: delayed intervention randomised controlled trial within the Medical Research Council (MRC) Framework to assess the effectiveness of a new palliative care service. BMC Palliat Care. 2006 Oct 2;5:7. doi: 10.1186/1472-684X-5-7. PMID 17014714
- [Result] Higginson IJ, Hart S, Burman R, Silber E, Saleem T, Edmonds P. Randomised controlled trial of a new palliative care service: Compliance, recruitment and completeness of follow-up. BMC Palliat Care. 2008 May 28;7:7. doi: 10.1186/1472-684X-7-7. PMID 18507817
- [Result] Higginson IJ, Hart S, Silber E, Burman R, Edmonds P. Symptom prevalence and severity in people severely affected by multiple sclerosis. J Palliat Care. 2006 Autumn;22(3):158-65. PMID 17058754
- [Derived] Higginson IJ, Costantini M, Silber E, Burman R, Edmonds P. Evaluation of a new model of short-term palliative care for people severely affected with multiple sclerosis: a randomised fast-track trial to test timing of referral and how long the effect is maintained. Postgrad Med J. 2011 Nov;87(1033):769-75. doi: 10.1136/postgradmedj-2011-130290. Epub 2011 Oct 6. PMID 21978993
- [Derived] Higginson IJ, McCrone P, Hart SR, Burman R, Silber E, Edmonds PM. Is short-term palliative care cost-effective in multiple sclerosis? A randomized phase II trial. J Pain Symptom Manage. 2009 Dec;38(6):816-26. doi: 10.1016/j.jpainsymman.2009.07.002. PMID 19833477
- See also: Overview of programme of studies in the department of palliative care of which this study is part — http://www.kcl.ac.uk/schools/medicine/depts/palliative/arp/eval/